CLINICAL TRIAL: NCT01677910
Title: A Phase 3, Randomized, Placebo-controlled, Parallel Group, Multicenter, Double-blind Study to Evaluate the Efficacy and Safety of Telotristat Etiprate (LX1606) in Patients With Carcinoid Syndrome Not Adequately Controlled by Somatostatin Analog (SSA) Therapy
Brief Title: TELESTAR (Telotristat Etiprate for Somatostatin Analogue Not Adequately Controlled Carcinoid Syndrome)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX1606.1-301-CS; LX1606.301 (Other: Lexicon Pharmaceuticals, Inc.); 2012-003460-47 (EudraCT Number)
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-01

CONDITIONS: Carcinoid Syndrome
MeSH Terms: conditions — Serotonin Syndrome | interventions — telotristat

STUDY DESIGN:
Intervention Model Description: Participants were randomized to one of three treatment arms in the double-blind treatment period. After completion of the double-blind treatment period, participants entered an open-label treatment period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 250 mg Telotristat Etiprate (Experimental): Following a 3 to 4-week run-in period on stable-dose somatostatin analog (SSA) therapy (octreotide or lanreotide) participants were randomized to receive one 250 mg telotristat etiprate tablet plus one placebo-matching telotristat etiprate tablet administered three times daily for 12 Weeks in the double-blind treatment period, followed by a 36 week open-label extension period.
  Interventions: Drug: Telotristat etiprate; Drug: Placebo-matching telotristat etiprate
- 500 mg Telotristat Etiprate (Experimental): Following a 3 to 4-week run-in period on stable-dose SSA therapy (octreotide or lanreotide) participants were randomized to receive, one telotristat etiprate 250 mg plus one placebo-matching telotristat etiprate tablet administered 3 times daily for 1 week, followed by two telotristat etiprate (250 mg) tablets administered three times daily for 11 weeks in the double-blind treatment period, followed by a 36 week open-label extension period.
  Interventions: Drug: Telotristat etiprate; Drug: Placebo-matching telotristat etiprate
- Placebo (Placebo Comparator): Following a 3 to 4-week run-in period on stable-dose SSA therapy (octreotide or lanreotide) participants were randomized to receive two placebo-matching telotristat etiprate tablets administered three times daily for 12 weeks in the double-blind treatment period, followed by a 36 week open-label extension period.
  Interventions: Drug: Placebo-matching telotristat etiprate
- Telotristat Etiprate Open-Label Extension (Experimental): Patients previously assigned to 250 mg or 500 mg three times daily of telotristat etiprate were administered two 250 mg telotristat etiprate tablets three times daily in a 36 week open-label extension (OLE) period. Patients previously assigned to placebo were administered one 250 mg telotristat etiprate tablet plus one placebo-matching tablet three times daily for one week, followed by two 250 mg telotristat etiprate tablets three times daily for 35 weeks.
  Interventions: Drug: Telotristat etiprate; Drug: Placebo-matching telotristat etiprate

INTERVENTIONS:
Drug: Telotristat etiprate — Telotristat etiprate tablets.
  Other Names: LX1606
  Arms: 250 mg Telotristat Etiprate; 500 mg Telotristat Etiprate; Telotristat Etiprate Open-Label Extension
Drug: Placebo-matching telotristat etiprate — Placebo-matching telotristat etiprate tablets.

SUMMARY:
The primary objective of the study is to confirm that at least 1 or more doses of telotristat etiprate compared to placebo is effective in reducing the number of daily bowel movements (BMs) from baseline averaged over the 12-week double-blind portion (Treatment Period) of the trial in patients not adequately controlled by current SSA therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically-confirmed, well-differentiated metastatic neuroendocrine tumor
* Documented history of carcinoid syndrome and currently experiencing ≥4 bowel movements per day during the Run-in period
* Currently receiving stable-dose somatostatin analog (SSA) therapy
* Minimum dose of long-acting release (LAR) or depot SSA therapy

  * Octreotide LAR at 30 mg every 4 weeks
  * Lanreotide Depot at 120 mg every 4 weeks
  * Patients who cannot tolerate SSA therapy at a level indicated above will be allowed to enter at their highest tolerated dose
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Presence of diarrhea attributed to any condition(s) other than carcinoid syndrome
* Karnofsky Performance status ≤60%
* Treatment with any tumor directed therapy, including interferon, chemotherapy, mechanistic target of rapamycin (mTOR) inhibitors <4 weeks prior to Screening, or hepatic embolization, radiotherapy, radiolabelled SSA, and/or tumor debulking <12 weeks prior to Screening
* History of short bowel syndrome (SBS)
* Clinically significant cardiac arrhythmia, bradycardia, tachycardia that would compromise patient safety or the outcome of the study
* Previous exposure to telotristat etiprate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2016-03-21 (Actual); Study Completion 2016-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Lapuerta, MD, Study Director — Lexicon Pharmaceuticals, Inc
Locations (69):
- United States (16):
  - Lexicon Investigational Site, Mobile, Alabama
  - Lexicon Investigational Site, Palo Alto, California
  - Lexicon Investigational Site, San Francisco, California
  - Lexicon Investigational Site, Orlando, Florida
  - Lexicon Investigational Site, Iowa City, Iowa
  - Lexicon Investigational Site, Lexington, Kentucky
  - Lexicon Investigational Site, Kenner, Louisiana
  - Lexicon Investigational Site, Boston, Massachusetts
  - Lexicon Investigational Site, Omaha, Nebraska
  - Lexicon Investigational Site, Buffalo, New York
  - Lexicon Investigational Site, New York, New York
  - Lexicon Investigational Site, Durham, North Carolina
  - Lexicon Investigational Site, Philadelphia, Pennsylvania
  - Lexicon Investigational Site, Fort Worth, Texas
  - Lexicon Investigational Site, Houston, Texas
  - Lexicon Investigational Site, McAllen, Texas
- Australia (6):
  - Lexicon Investigational Site, Kogara, New South Wales
  - Lexicon Investigational Site, Saint Leanoards, New South Wales
  - Lexicon Investigational Site, Herston, Queensland
  - Lexicon Investigational Site, Fitzroy, Victoria
  - Lexicon Investigational Site, Freemantle, Western Australia
  - Lexicon Investigational Site, Woodville South
- Belgium (3):
  - Lexicon Investigational Site, Edegem
  - Lexicon Investigational Site, Ghent
  - Lexicon Investigational Site, Yvoir
- Canada (2):
  - Lexicon Investigational Site, Calgary, Alberta
  - Lexicon Investigational Site, Halifax, Nova Scotia
- France (6):
  - Lexicon Investigational Site, Clichy
  - Lexicon Investigational Site, Lille
  - Lexicon Investigational Site, Lyon
  - Lexicon Investigational Site, Marseille
  - Lexicon Investigational Site, Strasbourg
  - Lexicon Investigational Site, Villejuif
- Germany (10):
  - Lexicon Investigational Site, Bad Berka
  - Lexicon Investigational Site, Berlin
  - Lexicon Investigational Site, Essen
  - Lexicon Investigational Site, Hamburg
  - Lexicon Investigational Site, Heidelberg
  - Lexicon Investigational Site, Lübeck
  - Lexicon Investigational Site, Mainz
  - Lexicon Investigational Site, Marburg
  - Lexicon Investigational Site, München
  - Lexicon Investigational Site, Neuss
- Lexicon Invetigational Site, Jerusalem, Israel
- Italy (9):
  - Lexicon Investigational Site, Bologna
  - Lexicon Investigational Site, Ferrara
  - Lexicon Investigational Site, Milan
  - Lexicon Investigational Site, Modena
  - Lexicon Investigational Site, Napoli
  - Lexicon Investigational Site, Orbassano
  - Lexicon Investigational Site, Perugia
  - Lexicon Investigational Site, Pisa
  - Lexicon Investigational Site, Rome
- Netherlands (4):
  - Lexicon Investigational Site, Amsterdam
  - Lexicon Investigational Site, Noord-Brahant
  - Lexicon Investigational Site, Noord-Holland
  - Lexicon Investigational Site, Zuid-Holland
- Spain (3):
  - Lexicon Investigational Site, Barcelona
  - Lexicon Investigational Site, Madrid
  - Lexicon Investigational Site, Seville
- Sweden (2):
  - Lexicon Investigational Site, Lund
  - Lexicon Investigational Site, Uppsala
- United Kingdom (7):
  - Lexicon Investigational Site, Basingstoke-Hampshire
  - Lexicon Investigational Site, Coventry
  - Lexicon Investigational Site, Glasgow
  - Lexicon Investigational Site, Headington-Oxford
  - Lexicon Investigational Site, London
  - Lexicon Investigational Site, Manchester
  - Lexicon Investigational Site, Newcastle upon Tyne

REFERENCES:
- [Derived] Srirajaskanthan R, Pavel M, Kulke M, Clement D, Houchard A, Keeber L, Weickert MO. Weight Maintenance up to 48 Weeks in Patients With Carcinoid Syndrome Treated With Telotristat Ethyl: Pooled Data From the Open-Label Extensions of the Phase III Clinical Trials TELESTAR and TELECAST. Clin Ther. 2021 Oct;43(10):1779-1785. doi: 10.1016/j.clinthera.2021.08.014. Epub 2021 Sep 28. PMID 34598813
- [Derived] Fust K, Maschio M, Kohli M, Singh S, Pritchard DM, Marteau F, Myrenfors P, Feuilly M. A Budget Impact Model of the Addition of Telotristat Ethyl Treatment to the Standard of Care in Patients with Uncontrolled Carcinoid Syndrome. Pharmacoeconomics. 2020 Jun;38(6):607-618. doi: 10.1007/s40273-020-00896-5. PMID 32157590
- [Derived] Dillon JS, Kulke MH, Horsch D, Anthony LB, Warner RRP, Bergsland E, Welin S, O'Dorisio TM, Kunz PL, McKee C, Lapuerta P, Banks P, Pavel M. Time to Sustained Improvement in Bowel Movement Frequency with Telotristat Ethyl: Analyses of Phase III Studies in Carcinoid Syndrome. J Gastrointest Cancer. 2021 Mar;52(1):212-221. doi: 10.1007/s12029-020-00375-2. PMID 32146619
- [Derived] Hudgens S, Ramage J, Kulke M, Bergsland E, Anthony L, Caplin M, Oberg K, Pavel M, Gable J, Banks P, Yang QM, Lapuerta P. Evaluation of meaningful change in bowel movement frequency for patients with carcinoid syndrome. J Patient Rep Outcomes. 2019 Oct 26;3(1):64. doi: 10.1186/s41687-019-0153-y. PMID 31655936
- [Derived] Cella D, Beaumont JL, Hudgens S, Marteau F, Feuilly M, Houchard A, Lapuerta P, Ramage J, Pavel M, Horsch D, Kulke MH. Relationship Between Symptoms and Health-related Quality-of-life Benefits in Patients With Carcinoid Syndrome: Post Hoc Analyses From TELESTAR. Clin Ther. 2018 Dec;40(12):2006-2020.e2. doi: 10.1016/j.clinthera.2018.10.008. Epub 2018 Nov 24. PMID 30477789
- [Derived] Weickert MO, Kaltsas G, Horsch D, Lapuerta P, Pavel M, Valle JW, Caplin ME, Bergsland E, Kunz PL, Anthony LB, Grande E, Oberg K, Welin S, Lombard-Bohas C, Ramage JK, Kittur A, Yang QM, Kulke MH. Changes in Weight Associated With Telotristat Ethyl in the Treatment of Carcinoid Syndrome. Clin Ther. 2018 Jun;40(6):952-962.e2. doi: 10.1016/j.clinthera.2018.04.006. Epub 2018 May 1. PMID 29724499

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 48 investigative sites in Australia, Belgium, Canada, France, Germany, Israel, Italy, Netherlands, Spain, Sweden, United Kingdom, and the United States from 08 January 2013 to 21 March 2016.
Pre-assignment Details: Patients with Carcinoid Syndrome not adequately controlled by somatostatin analog (SSA) therapy were assigned in a 1:1:1 ratio to receive placebo, 250 mg or 500 mg telotristat etiprate (LX1606) in the double-blind period and were eligible to receive 500 mg telotristat etiprate in the 36 week open-label extension. 136 randomized;1 patient twice.
Period: Double-Blind Treatment Period
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate | Telotristat Etiprate Open-Label Extension
Started | 45 | 45 | 45 | 0
Completed | 38 | 42 | 38 | 0
Not Completed | 7 | 3 | 7 | 0
Not completed — Adverse Event | 6 | 2 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal of consent | 1 | 0 | 3 | 0
Not completed — Reason Not Specified | 0 | 1 | 0 | 0
Period: Open-Label Extension Period (OLE)
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate | Telotristat Etiprate Open-Label Extension
Started | 0 | 0 | 0 | 115
Completed | 0 | 0 | 0 | 79
Not Completed | 0 | 0 | 0 | 36
Not completed — Physician Decision | 0 | 0 | 0 | 4
Not completed — Reason not Specified | 0 | 0 | 0 | 2
Not completed — Withdrawal of Consent | 0 | 0 | 0 | 9
Not completed — Lack of Efficacy | 0 | 0 | 0 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 15
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate | Total
Number analyzed (Participants) | 45 | 45 | 45 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (8.67) | 62.4 (9.12) | 64.9 (9.06) | 63.2 (9.28)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 25 | 26 | 22 | 73
  ≥ 65 years | 20 | 19 | 23 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 20 | 65
  Male | 24 | 21 | 25 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity data was not provided for 1 participant in France.
  Participants
    Hispanic or Latino | 0 | 0 | 1 | 1
    Not Hispanic or Latino | 45 | 44 | 44 | 133
    Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race information was not provided for 11 participants from France.
  Participants
    American Indian or Alaska Native | 1 | 0 | 0 | 1
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 1 | 0 | 0 | 1
    White | 40 | 41 | 40 | 121
    More than one race | 0 | 0 | 1 | 1
    Unknown or Not Reported | 3 | 4 | 4 | 11
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 2 | 2 | 7
  Sweden | 3 | 3 | 3 | 9
  Netherlands | 2 | 3 | 3 | 8
  Belgium | 1 | 0 | 0 | 1
  United States | 12 | 13 | 12 | 37
  United Kingdom | 8 | 3 | 8 | 19
  Italy | 1 | 4 | 3 | 8
  Israel | 2 | 0 | 0 | 2
  Australia | 1 | 2 | 3 | 6
  France | 3 | 4 | 4 | 11
  Germany | 5 | 8 | 6 | 19
  Spain | 4 | 3 | 1 | 8
Somatostatin Analog (SSA) Therapy Schedule at Study Entry [Count of Participants; unit: Participants] — Patients who were on a 2-week SSA therapy or receiving SSA therapy via a subcutaneous continuous infusion pump are included in the "4-week" category.
  Participants
    3-Week | 11 | 11 | 17 | 39
    4-Week | 34 | 34 | 28 | 96
SSA Therapy Name at Study Entry [Count of Participants; unit: Participants]
  Octreotide | 30 | 40 | 33 | 103
  Lanreotide | 15 | 5 | 12 | 32
Childbearing Potential [Count of Participants; unit: Participants]
  Yes | 3 | 0 | 0 | 3
  No | 18 | 24 | 20 | 62
  Not Applicable | 24 | 21 | 25 | 70
Urinary 5-hydroxyindoleacetic acid (u5-HIAA) at Randomization [Count of Participants; unit: Participants] — ULN=upper limit of normal
  Participants
    ≤ULN | 12 | 12 | 12 | 36
    >ULN | 26 | 26 | 26 | 78
    Unknown | 7 | 7 | 7 | 21
Region [Count of Participants; unit: Participants] — North America includes USA and Canada; Europe includes Belgium, France, Germany, Italy, Netherlands, Spain, Sweden, and United Kingdom; Rest of the World includes Australia and Israel.
  Participants
    North America | 15 | 15 | 14 | 44
    Europe | 27 | 28 | 28 | 83
    Rest of the World | 3 | 2 | 3 | 8
Weight [Mean (Standard Deviation); unit: kilogram (kg)] — Population: Weight data was not available for all participants.
  kilogram (kg)
    number analyzed (Participants) | 43 | 44 | 44 | 131
    (all) | 70.87 (13.940) | 70.05 (14.832) | 73.44 (19.971) | 71.46 (16.419)
Height [Mean (Standard Deviation); unit: centimeter (cm)] — Population: Height data was not available for all participants.
  centimeter (cm)
    number analyzed (Participants) | 39 | 41 | 40 | 120
    (all) | 168.8 (10.707) | 169.32 (9.607) | 169.93 (10.436) | 169.35 (10.175)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI was calculated by weight (kg) / (height (cm) *0.01)^2. Population: Not all participants had weight and height data available to calculate BMI.
  kg/m^2
    number analyzed (Participants) | 38 | 41 | 39 | 118
    (all) | 25.13 (4.790) | 24.26 (4.702) | 25.24 (5.352) | 24.87 (4.931)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Number of Bowel Movements (BMs) Per Day Averaged Over 12 Weeks
Description: Participants recorded the number of bowel movements per day in a daily diary. The total number of BMs per day were averaged over the 12-week period. A negative change from Baseline indicates improvement.
Time Frame: Baseline and 12 Weeks
Population: Participants from the Intent-to-treat population, all randomized participants, with data available were included in the analyses.
Measure: Mean (Standard Deviation); unit: counts/day
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate
Number analyzed (Participants) | 45 | 45 | 45
counts/day | -0.623 (0.8275) | -1.433 (1.3652) | -1.455 (1.3098)
Statistical Analysis 1: Comparison: Placebo vs 250 mg Telotristat Etiprate; Primary analysis used a blocked 2-sample Wilcoxon rank sum statistic stratified by the urinary 5-HIAA stratification at randomization; Test type: Superiority; p < 0.001, Wilcoxon rank sum; Mean Difference (Net) = -0.81, 95% CI 2-sided [-1.283 to -0.337] — Mean difference is calculated as LX1606-Placebo
Statistical Analysis 2: Comparison: Placebo vs 500 mg Telotristat Etiprate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Wilcoxon rank sum; Mean Difference (Net) = -0.833, 95% CI 2-sided [-1.292 to -0.374] — Mean difference is calculated as LX1606-Placebo

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) in the Double-Blind Treatment Period
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A TEAE was an AE reported after the first dose of randomized treatment on Day 1.
Time Frame: First dose of study drug to within 30 days of last dose of study drug in the Double-Blind Treatment Period (Up to 17.6 Weeks)
Population: Safety population, defined as all subjects who received at least one dose of study drug was used for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate
Number analyzed (Participants) | 45 | 45 | 45
Participants | 39 | 37 | 42

3. Secondary Outcome: Change From Baseline in Urinary 5-hydroxyindoleacetic Acid (u5-HIAA) Levels
Description: u5-HIAA is a standard test used in clinical practice to assess neuroendocrine tumor (NET) activity and is collected as a 24-hour urine specimen. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: Participants from the Intent-to-treat population, all randomized participants, with u5-HIAA data available at Baseline and Week 12 were included in the analyses.
Measure: Mean (Standard Deviation); unit: mg/24 hours
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate
Number analyzed (Participants) | 30 | 32 | 31
mg/24 hours | 11.350 (35.0346) | -40.134 (84.7663) | -57.519 (82.3273)

4. Secondary Outcome: Change From Baseline in the Number of Daily Cutaneous Flushing Episodes Averaged Across All Time-Points
Description: Participants recorded the number daily flushing episodes per day in a daily diary. The total number of flushing episodes per day were averaged over the 12-week period. A negative change from Baseline indicates improvement.
Time Frame: Baseline and 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: counts/day
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate
Number analyzed (Participants) | 45 | 45 | 45
counts/day | -0.164 (1.1572) | -0.296 (1.3097) | -0.525 (1.3413)

5. Secondary Outcome: Change From Baseline in Abdominal Pain Averaged Across All Time-Points
Description: Participants recorded abdominal pain in a daily diary. Participants evaluated the level of any abdominal pain using an 11-point numeric rating scale, where: 0=no pain to 10=worst pain ever experienced. The average daily abdominal pain was averaged over the 12-week period. A negative change from Baseline indicates improvement.
Time Frame: Baseline and 12 Weeks
Population: Participants from the Intent-to-treat population, all randomized participants, with available data were included in the analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate
Number analyzed (Participants) | 45 | 45 | 45
units on a scale | -0.226 (1.1601) | -0.489 (1.4423) | -0.333 (1.1784)

6. Primary Outcome: Number of Participants With TEAEs in the Open-Label Extension Period
Description: as for outcome 2
Time Frame: First dose of study drug to within 30 days of last dose of study drug in the Open-Label Extension Period (Up to 54.3 Weeks)
Population: Safety population, defined as all subjects who received at least one dose of study drug was used for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Telotristat Etiprate Open-Label Extension
Number analyzed (Participants) | 115
Participants | 110

ADVERSE EVENTS:
Time Frame: First dose of study drug to within 30 days of last dose of study drug (Up to 72.2 Weeks)
Groups:
- Placebo: Following a 3 to 4-week run-in period on stable-dose SSA therapy (octreotide or lanreotide) participants were randomized to receive two placebo-matching telotristat etiprate tablets administered three times daily for 12 weeks in the double-blind treatment period.
- 250 mg Telotristat Etiprate: Following a 3 to 4-week run-in period on stable-dose somatostatin analog (SSA) therapy (octreotide or lanreotide) participants were randomized to receive one 250 mg telotristat etiprate tablet plus one placebo-matching telotristat etiprate tablet administered three times daily for 12 Weeks in the double-blind treatment period.
- 500 mg Telotristat Etiprate: Following a 3 to 4-week run-in period on stable-dose SSA therapy (octreotide or lanreotide) participants were randomized to receive, one 250 mg telotristat etiprate tablet plus one placebo-matching telotristat etiprate tablet administered 3 times daily for 1 week, followed by two 250 mg telotristat etiprate tablets administered three times daily for 11 weeks in the double-blind treatment period.
Arm/Group | Placebo | 250 mg Telotristat Etiprate | 500 mg Telotristat Etiprate | Telotristat Etiprate Open-Label Extension
All-Cause Mortality (participants affected / at risk) | 3/45 | 1/45 | 1/45 | 9/115
Serious Adverse Events (participants affected / at risk) | 7/45 | 7/45 | 8/45 | 37/115
Other Adverse Events (participants affected / at risk) | 39/45 | 37/45 | 42/45 | 110/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=45) | 250 mg Telotristat Etiprate (N=45) | 500 mg Telotristat Etiprate (N=45) | Telotristat Etiprate Open-Label Extension (N=115)
Desseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Carcinoid heart disease (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 0 | 0
Carcinoid syndrome (Endocrine disorders) | 0 | 0 | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 5
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Disease progression (General disorders) | 1 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Investigation (Investigations) | 0 | 2 | 1 | 4
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Pancreatic neuroendocrine tumor metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Skin neoplasm excision (Surgical and medical procedures) | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 1
Radiotherapy (Surgical and medical procedures) | 0 | 0 | 0 | 3
Chemotherapy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Gastrostomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Nephrostomy tube placement (Surgical and medical procedures) | 0 | 0 | 0 | 1
Surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1
Therapeutic embolisation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 3
Fatigue (General disorders) | 0 | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post embolisation syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1
Cholangiogram (Investigations) | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Peritoneal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colonic stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 2
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Pyonephrosis (Infections and infestations) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=45) | 250 mg Telotristat Etiprate (N=45) | 500 mg Telotristat Etiprate (N=45) | Telotristat Etiprate Open-Label Extension (N=115)
Nausea (Gastrointestinal disorders) | 5 | 6 | 14 | 27
Abdominal pain (Gastrointestinal disorders) | 8 | 5 | 10 | 35
Vomiting (Gastrointestinal disorders) | 4 | 2 | 5 | 16
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 5 | 13
Abdominal distension (Gastrointestinal disorders) | 3 | 2 | 1 | 13
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 0 | 11
Flatulence (Gastrointestinal disorders) | 1 | 3 | 2 | 11
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 1 | 0
Fatigue (General disorders) | 4 | 4 | 7 | 13
Asthenia (General disorders) | 3 | 2 | 1 | 11
Oedema peripheral (General disorders) | 2 | 3 | 2 | 10
Nasopharyngitis (Infections and infestations) | 1 | 2 | 3 | 6
Pneumonia (Infections and infestations) | 0 | 0 | 3 | 0
Gamma-glutamyl transferase increased (Investigations) | 0 | 4 | 4 | 9
Alanine amino transferase increased (Investigations) | 0 | 1 | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 7 | 13
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 3 | 5 | 8
Headache (Nervous system disorders) | 2 | 5 | 5 | 12
Dizziness (Nervous system disorders) | 2 | 0 | 4 | 0
Memory impairment (Nervous system disorders) | 3 | 0 | 1 | 0
Depression (Psychiatric disorders) | 3 | 2 | 7 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Flushing (Vascular disorders) | 2 | 3 | 3 | 7
Hypertension (Vascular disorders) | 0 | 0 | 0 | 6
General physical health deterioration (General disorders) | 0 | 0 | 0 | 8
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 9
Decreased interest (Psychiatric disorders) | 0 | 0 | 0 | 7
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 6
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 8
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 10
Pyrexia (General disorders) | 2 | 3 | 0 | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 6
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least thirty (30) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any confidential information, proprietary information, or patentable subject matter.